CLINICAL TRIAL: NCT00000337
Title: Infusion Laboratory: Protocol 1 - Selegeline
Brief Title: Infusion Laboratory: Protocol 1 - Selegeline - 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-3-0010-2; Y01-3-0010-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1996-08

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Selegiline

INTERVENTIONS:
Drug: Selegiline

SUMMARY:
The purpose of this study is to determine the effects of selegiline on the subjective and physiological effects of cocaine challenge in chronic crack abusers, and to evaluate clinical safety issues pertaining to selegeline, to cocaine and their interaction in a chronic crack dependent population.

DETAILED DESCRIPTION:
To develop a medication for the treatment of cocaine addiction using a medical human physio-neuro-psycho-immunology laboratory setting. To characterize this cocaine abusing population on a variety of psychological and physicologically measures over time from withdrawal through pere and post cocaine administration. To determine the effects of selegeline on the subjective and physiological effects of cocaine challenge in chronic crack abusers. To evaluate clinical safety issues pertaining to selegeline, to cocaine and their interaction in a chronic crack dependent population.

ELIGIBILITY:
Inclusion Criteria:

M/F, ages 21-50. Meet DSM-IV criteria for cocaine dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nuring women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical condtions that deem participation to be unsafe.

Ages: 31 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-11

PRIMARY OUTCOMES:
Degree of drug craving
History, incidence and amount of drug use
Type and severity of stimulant withdrawal symptoms
Population incidence of symptoms of depression, possible organic brain syndrome deficits
Frequency and intensity of drug use and sexual behaviors at risk for HIV
Evidence of change in neurophysiology and brain activity
Evidence of change in subjective responses to cocaine challenge
Clinical physiological response to cocaine challenge - especially adverse effects measures
Degree to which study medication influences changes in #6, 7 & 8 above (possible efficacy measure)
Characterization of study population

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States

REFERENCES:
- [Background] 1996 CPDD: "Acute cocaine administration reverses EEG signs of cocaine withdrawal.". 1996 CPDD: "Acute cocaine administration reverses EEG signs of cocaine withdrawal."